CLINICAL TRIAL: NCT00541190
Title: Absorptive Clearance in the Cystic Fibrosis Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Tim Corcoran, Assistant Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO07060240; NIH K25 HL081533-02
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Results first posted 2012-02-03 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; mucociliary clearance; outcome measures
MeSH Terms: conditions — Cystic Fibrosis | interventions — Technetium; Indium; Indium-111; Pentetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cystic fibrosis (Experimental): Cystic fibrosis patients
  Interventions: Other: Technetium [Tc-99m] sulfur colloid and Indium [In-111] DTPA
- healthy controls (Experimental): Healthy control subjects
  Interventions: Other: Technetium [Tc-99m] sulfur colloid and Indium [In-111] DTPA

INTERVENTIONS:
Other: Technetium [Tc-99m] sulfur colloid and Indium [In-111] DTPA — Subjects perform a single nuclear medicine scan after inhaling an aerosol containing Technetium 99m sulfur colloid and Indium 111 DTPA.

SUMMARY:
The objective of this overall project is to develop a new aerosol-based technique for quantifying liquid absorption in the airways of subjects with cystic fibrosis(CF) that can be used to help develop new therapies. In CF, mutations in the CF gene result in dysfunction of the Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) ion channel on the cells that line the airway epithelium, causing improper fluxes of ions such as sodium, chloride, and bicarbonate. The so called "low volume" hypothesis of CF pathogenesis contends that abnormal absorption of ions from the airways causes excessive absorption of liquid, resulting in an airway surface liquid layer that is dehydrated and difficult to clear. Here we are measuring the absorption rate of a radiolabeled small molecule (DTPA) from the lungs of cystic fibrosis patients and healthy controls. We hypothesize that the molecule will absorb more quickly in cystic fibrosis patients. Further studies will be performed to determine if DTPA absorption is related to liquid absorption in the airways.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis subjects and healthy controls
* Age ≥ 18 years
* Diagnosis of cystic fibrosis as determined by sweat test or genotype and clinical symptoms (CF subjects)
* Clinically stable as determined by the investigator (pulmonologist)

Exclusion Criteria:

* Reactive airways disease
* Tobacco smokers (regular smoking within 6 months of enrollment)
* Positive urine pregnancy test on the day of testing
* FEV1p value of < 50%
* SaO2 < 92%, or if they require supplemental oxygen.
* Subjects performing other radioisotope studies within the last 2 weeks will be excluded.
* Healthy subjects with any history of lung disease will be excluded.
* Women currently breastfeeding
* Subjects not willing to stop treatments with inhaled hypertonic saline for 48 hours in advance of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy E Corcoran, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Locke LW, Myerburg MM, Weiner DJ, Markovetz MR, Parker RS, Muthukrishnan A, Weber L, Czachowski MR, Lacy RT, Pilewski JM, Corcoran TE. Pseudomonas infection and mucociliary and absorptive clearance in the cystic fibrosis lung. Eur Respir J. 2016 May;47(5):1392-401. doi: 10.1183/13993003.01880-2015. Epub 2016 Mar 23. PMID 27009167
- [Derived] Corcoran TE, Thomas KM, Myerburg MM, Muthukrishnan A, Weber L, Frizzell R, Pilewski JM. Absorptive clearance of DTPA as an aerosol-based biomarker in the cystic fibrosis airway. Eur Respir J. 2010 Apr;35(4):781-6. doi: 10.1183/09031936.00059009. Epub 2009 Aug 28. PMID 19717485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cystic fibrosis subjects were recruited during normal clinical visits. Healthy control subjects were recruited using posted advertisement.
Pre-assignment Details: All enrolled subjects performed a single nuclear medicine imaging study.
Groups:
- Healthy Controls: Healthy subjects.
Period: Overall Study
Arm/Group | Cystic Fibrosis | Healthy Controls
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cystic Fibrosis | Healthy Controls | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (11) | 29 (7) | 29 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Absorptive Clearance Rate
Description: The absorptive clearance rate is the percentage of the radiolabeled small molecule DTPA that is cleared through absorption over a 60 minute period. Total DTPA clearance includes absorptive and mucociliary components. The mucociliary component is determined by measuring the clearance of a radiolabeled particle over the same period (Technetium 99m sulfur colloid; Tc-SC), and subtracted from total DTPA clearance in order to determine the absorptive component. Here we specifically report absorption from the central lung zone to capture the behavior within the airways.
Time Frame: single measurement
Population: No formal power analysis was performed for this pilot study. Two subjects (one CF, one control) were identified as obvious outliers with whole lung Tc-SC clearance rates more than two standard deviations above the average of the group. These outliers were excluded from further analyses.
Measure: Mean (Standard Deviation); unit: percentage of DTPA absoprtion per hour
Groups:
- Cystic Fibrosis: Cystic fibrosis patients - subjects inhaled a nebulized mixture of Indium 111 DTPA and Technetium 99m sulfur colloid.
- Healthy Controls: Healthy subjects without lung disease - subjects inhaled a nebulized mixture of Indium 111 DTPA and Technetium 99m sulfur colloid.
Arm/Group | Cystic Fibrosis | Healthy Controls
Number analyzed (Participants) | 9 | 10
percentage of DTPA absoprtion per hour | 42 (11) | 32 (7)

2. Secondary Outcome: Mucociliary Clearance Rate
Description: Mucociliary clearance rate represents the rate at which the lungs clear an inhaled particulate. Here it specifically represents the percentage of inhaled Technetium 99m sulfur colloid cleared from the lungs over a 60 minute period. This is reported based on "whole lung" areas to allow comparisons with previous studies.
Time Frame: single measurement
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage lung clearance per hour
Arm/Group | Cystic Fibrosis | Healthy Controls
Number analyzed (Participants) | 9 | 10
percentage lung clearance per hour | 8 (4) | 7 (4)

ADVERSE EVENTS:
Arm/Group | Cystic Fibrosis | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No